CLINICAL TRIAL: NCT02037854
Title: PEP-1324: Glycemic Response Testing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1324
Record Dates: First submitted 2014-01-13; First posted 2014-01-16 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Glycemic Response

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): A nutrient formulation without the active ingredient
  Interventions: Other: Nutrient formulation
- Nutrient formulation (Experimental): Nutrient formulations with variable amounts of active ingredients.
  Interventions: Other: Nutrient formulation

INTERVENTIONS:
Other: Nutrient formulation

SUMMARY:
The purpose of this study is to assess whether food ingredient(s) affect glycemic and insulinemic responses.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-75 years of age
* Subject is male or non-pregnant females, 18-75 years of age, inclusive
* Subject has a body mass index (BMI) ≥ 20.0 and < 35 kg/m² at screening (visit 1).
* Subject has to be non-smoker.
* Subject is willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
* Subject is willing to maintain current dietary supplement use throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the GI labs. Failure to comply will result in a rescheduled test visit.
* Subject has normal fasting serum glucose (<7.0mmol/L capillary corresponding to whole blood glucose <6.3mmol/L).
* Subject is willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits.
* Subject has no health conditions that would prevent him from fulfilling the study requirements as judged by the Investigator on the basis of medical history.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incremental area under the blood glucose response cruve | 0-2 hours

SECONDARY OUTCOMES:
peak blood glucose | 0-2 hours
peak insulin | 0-2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- GI Labs, Toronto, Ontario, Canada